CLINICAL TRIAL: NCT06683508
Title: A Phase 2, Parallel-Group, Double-Blind Study to Investigate Weight Management With LY3549492 Once Daily Compared With Placebo in Adult Participants With Obesity or Overweight
Brief Title: A Study to Investigate Weight Management With LY3549492 Compared With Placebo in Adult Participants With Obesity or Overweight
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27240; W8M-MC-GN01 (Other: Eli Lilly and Company); W8M-MC-CWMM (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3549492 Dose 1 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 2 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 3 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 4 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- LY3549492 Dose 5 (Experimental): Participants will receive LY3549492 orally
  Interventions: Drug: LY3549492
- Placebo (Placebo Comparator): Participants will receive Placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3549492 — Administered orally
  Arms: LY3549492 Dose 1; LY3549492 Dose 2; LY3549492 Dose 3; LY3549492 Dose 4; LY3549492 Dose 5
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study, performed under the master protocol W8M-MC-CWMM (NCT06143956), is to evaluate the effects of LY3549492 in adults with obesity or overweight. Participation in the study will last about one year.

ELIGIBILITY:
Inclusion Criteria:

W8M-MC-GN01:

* Assigned male at birth
* Assigned female at birth, who are of non-childbearing potential

W8M-MC-CWMM:

* Have a BMI of

  * ≥ 30 kilograms per square meter (kg/m²) or
  * ≥ 27 kg/m² and < 30 kg/m² with at least one weight-related comorbidity
* Have had a stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss)

Exclusion Criteria:

W8M-MC-GN01:

* Have Type 2 Diabetes Mellitus or Type 1 Diabetes Mellitus
* Have a history of acute or chronic pancreatitis
* Have renal impairment
* Individuals who are of childbearing potential

W8M-MC-CWMM:

* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening.
* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults, or history of ketoacidosis or hyperosmolar coma.
* Have poorly controlled hypertension.
* Have signs and symptoms of any liver disease other than nonalcoholic fatty liver disease.
* Have any of the following cardiovascular conditions within 3 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure.
* Have a history of symptomatic gallbladder disease within the past 2 years
* Have a lifetime history of suicide attempts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 36

SECONDARY OUTCOMES:
Change from Baseline in Body Weight (kilograms) | Baseline, Week 36
Percentage of Participants who Achieve ≥5% Body Weight Reduction | Baseline, Week 36
Percentage of Participants who Achieve ≥10% Body Weight Reduction | Baseline, Week 36
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 36
Pharmacokinetics (PK): Average Concentration of LY3549492 | Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (49):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson, Tucson, Arizona
  - NorCal Medical Research, Inc, Greenbrae, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Medical Research Partners, Ammon, Idaho
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Knownwell, Needham, Massachusetts
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Medication Management, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Quality Medical Research, Nashville, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study to Investigate Weight Management with LY3549492 Compared with Placebo in Adult Participants With Obesity or Overweight — https://trials.lilly.com/en-US/trial/554575